CLINICAL TRIAL: NCT06223737
Title: Characterization of Patients Suffering From Adult Spine Deformities With Optoelectronic Motion Analysis
Brief Title: Spine Deformity Patients With Optoelectronic Motion Capture
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Schulthess Klinik (Other)
Collaborators: ETH Zurich (Other); Bern University of Applied Sciences (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Factorial | Masking: None | Purpose: Screening
Other Study IDs: SHPL_Def_00782
Record Dates: First submitted 2023-09-05; First posted 2024-01-25 (Actual); Last update posted 2024-11-29 (Actual); Status verified 2024-11

CONDITIONS: Spine Deformity
Keywords: Adult Spine Deformity; Surgical Planning; Spinal Deformity; Optoelectronic Motion Analysis; Biplanar Radiography; Absolute Spinal Curvature
MeSH Terms: interventions — Motion Capture

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- patients non-operated (Active Comparator): Each patient will be measured for an EOS x-ray and at the human performance lab at the clinic for optoelectronic motion capture of the spinal movements.
  Interventions: Diagnostic Test: EOS x-ray; Diagnostic Test: Motion capture
- patients operated (Active Comparator): Each patient will be measured for an EOS x-ray and at the human performance lab at the clinic for optoelectronic motion capture of the spinal movement
  Interventions: Diagnostic Test: EOS x-ray; Diagnostic Test: Motion capture
- healthy controls (Other): Each participant will be measured as control group for an EOS x-ray and at the human performance lab at the clinic for optoelectronic motion capture of the spinal movement
  Interventions: Diagnostic Test: EOS x-ray; Diagnostic Test: Motion capture

INTERVENTIONS:
Diagnostic Test: EOS x-ray — After marking the anatomical landmarks where later on skin markers will be placed, radiopaque markers are attached for the radiographic examination with the EOS system. Images are taken from the positions standing and sitting
Diagnostic Test: Motion capture — The used marker set is the IfB marker set (List et al. 2013), consisting of 40 skin markers on the lower extremities, 7 on the pelvis, 24 on the trunk and 6 on the upper extremities. For the later musculoskeletal modelling the IfB marker set is extended with 7 additional markers on the spinal thoracic processes. All markers will be placed by skilled operators.
  The test procedure consists of six trials, namely a standing trial in an anatomic upright position and a calibration motion as well as four basic motion tasks to define functional estimated joint axis, respectively centers (each performed twice).
  Tasks: standing, maximal flexion-extension, lateral bending, axial rotation, lifting, holding load, walking, step up, sitting and sit-to-stand
  Other Names: Optoelectronic camera system

SUMMARY:
Aging-induced changes in the spine can lead to adult spinal deformity, causing a forward and/or lateral shift of the trunk. While mild cases may have compensatory mechanisms, severe deformities necessitate treatment. Surgery with instrumentation effectively corrects deformities, but complications are common. Precise pre-operative planning based on X-rays is essential. However, radiological imaging has limitations, including ionizing radiation exposure and static nature. Marker-based optoelectronic motion analysis systems offer potential benefits for dynamic spine assessment.

This study aims to test the feasibility of using motion analysis systems to characterize spinal alignment and balance in patients with adult spine deformity. The primary objective is to assess the practical implementation, measurement capability, and resources required for motion analysis. Secondary objectives include investigating errors in absolute spinal curvature assessment and developing compensation strategies.

The project will recruit 20 patients (non-operated and operated) seeking medical attention for adult spine deformities and 10 healthy controls. Participants will undergo biplanar imaging and motion analysis to capture static and dynamic spine alignment during common activities. The data will help build patient-specific musculoskeletal models, offering potential insights into improving surgical planning for adult spine deformities.

DETAILED DESCRIPTION:
Aging and degeneration can lead to changes in the spine, causing adult spinal deformities like loss of lumbar lordosis, thoracic hyperkyphosis, and scoliosis. Severe deformities can be highly debilitating, necessitating treatments. Surgery using instrumentation, such as pedicle screws, rods, and cages, can effectively correct adult spine deformities. However, complications and failures are common.

Precise pre-operative planning based on standing X-rays is crucial before attempting correction. Radiographic parameters, including pelvic incidence (PI), sagittal vertical axis (SVA), lumbar lordosis, thoracic kyphosis, coronal Cobb angles, and vertebral rotation, are measured to evaluate the patient's standing posture and compensatory mechanisms.

Limitations in traditional radiological imaging for spinal alignment assessment include ionizing radiation exposure and lack of information on dynamic spine responses during various activities. To address these limitations, marker-based optoelectronic motion analysis systems have been proposed to characterize dynamic spinal alignment and movement during different activities. This technology has shown promise in assessing spinal curvature changes reliably.

This research aims to investigate the feasibility of using optoelectronic motion analysis systems to characterize spinal alignment and balance in patients with adult spine deformity. The primary objective is to assess the practical implementation, measurement capability, and resources required for motion analysis. Secondary objectives include exploring potential strategies to compensate for errors in absolute spinal curvature assessment due to markers on soft tissue.

The study will recruit 20 patients seeking medical attention for adult spine deformities (divided into non-operated and operated subgroups) and 10 healthy controls. Participants will undergo biplanar imaging and motion analysis to capture static and dynamic spine alignment during various activities. The data obtained will be used to build patient-specific musculoskeletal models, offering potential insights into improving surgical planning for adult spine deformities.

The findings of this study may lead to advancements in understanding spinal deformities and help in developing personalized treatment strategies to improve outcomes for patients suffering from adult spine deformities.

ELIGIBILITY:
Inclusion Criteria:

* both male and female subjects
* BMI < 30 kg/m2
* cognitively intact
* degenerative spinal deformity presenting with at least one criterion:

  * Coronal Cobb angle ≥20°
  * sagittal vertical axis (SVA) ≥5 cm
  * thoracic kyphosis (TK) ≥60°
  * pelvic tilt (PT) ≥25°.

Exclusion Criteria:

* age under 18 years or over 75 years
* any prior spinal surgery or other musculoskeletal surgery having an impact on movement
* pregnancy
* inability to perform the planned set of daily activities
* inability to give consent.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-05-01 (Estimated); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Feasibility of using motion analysis systems to characterize spinal alignment and balance in static and dynamic conditions | 1-2hours
  This primary outcome investigation focuses on assessing key spinal parameters, including lumbar lordosis, pelvic tilt, thoracic kyphosis, and the severity of scoliosis, in static conditions. Additionally, the study captures the same variables during the performance of common daily activities, such as gait, maximal flexion, trunk torsion, lifting loads, walking with loads, and sit-to-stand transitions. The goal is to understand the feasibility of using optoelectronic motion analysis to provide comprehensive insights into spinal alignment and balance for both operated and non-operated adult spine deformity patients.

SECONDARY OUTCOMES:
investigate and quantify the well-known errors in the assessment of the absolute spinal curvature | 1-2hours
  The secondary outcome investigation focuses on exploring and quantifying known errors associated with the assessment of absolute spinal curvature, particularly when soft tissue markers are employed. The study aims to develop strategies to compensate for these errors, considering the challenges posed by attaching markers on top of soft tissues. The objective is to enhance the accuracy of spinal curvature measurements obtained through optoelectronic motion analysis, contributing to improved surgical planning for adult spine deformity cases.

CONTACTS AND LOCATIONS:
Locations (1):
- Schulthess Klinik, Zurich, Switzerland